CLINICAL TRIAL: NCT00674973
Title: A Phase II Biomarker Identification Trial for Erlotinib (Tarceva®) in Patients With Advanced Pancreatic Carcinoma
Brief Title: A Biomarker Identification Trial of Tarceva (Erlotinib) in Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BO21129; 2007-003738-40 (EudraCT Number)
Record Dates: First submitted 2008-04-30; First posted 2008-05-08 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Erlotinib (Experimental): Participants with advanced pancreatic carcinoma with Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 to 2, who had failed 1 prior regimen of chemotherapy or who were considered unsuitable for chemotherapy, received erlotinib 150 mg orally once daily until disease progression, unacceptable toxicity, withdrawal, or death.
  Interventions: Drug: Erlotinib
- Placebo (Placebo Comparator): Participants with advanced pancreatic carcinoma with ECOG PS score of 0 to 2, who had failed 1 prior regimen of chemotherapy or who were considered unsuitable for chemotherapy, received placebo matching to erlotinib 150 mg tablet orally once daily until disease progression, unacceptable toxicity, withdrawal, or death.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erlotinib — Participants received erlotinib 150 mg tablet orally once daily.
  Other Names: Tarceva
  Arms: Erlotinib
Drug: Placebo — Participants received placebo matching to erlotinib 150 mg tablet orally once daily.
  Arms: Placebo

SUMMARY:
This study is designed to identify biomarkers which may predict improvement in progression free survival from treatment with Tarceva, in patients with advanced pancreatic cancer who failed one prior regimen of standard chemotherapy or who are deemed unsuitable for chemotherapy. It will also assess the efficacy and safety of Tarceva in this patient population. Patients will be randomized to receive either Tarceva 150mg/day po, or placebo po daily. Tumor tissue will be used for biomarker analysis. The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* histologically or cytologically documented locally advanced-unresectable or metastatic pancreatic cancer;
* measurable disease according to RECIST;
* failure of at least one prior chemotherapy regimen, or who are deemed unsuitable for chemotherapy;
* ECOG performance status of 0-2.

Exclusion Criteria:

* local or locally advanced-resectable pancreatic cancer;
* any other malignancies within last 5 years, except for adequately treated cancer in situ of the cervix, or basal or squamous cell skin cancer;
* major surgery within 2 weeks prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (60):
- Australia (4):
  - Kogarah, New South Wales
  - St Leonards, New South Wales
  - Sydney, New South Wales
  - Box Hill, Victoria
- Brazil (7):
  - Salvador, Bahia, Estado de Bahia
  - Belo Horizonte, Minas Gerais
  - Curitiba, Paraná
  - Ijuí, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Jaú, São Paulo
  - São Paulo, São Paulo
- Bulgaria (5):
  - Gabrovo
  - Pleven
  - Plovdiv
  - Sofia
  - Vratsa
- Zagreb, Croatia
- Germany (8):
  - Bochum
  - Cologne
  - Dresden
  - Esslingen am Neckar
  - Greifswald
  - Hamburg
  - Saarbrücken
  - Ulm
- Hong Kong, Hong Kong
- India (10):
  - Bangalore
  - Chennai
  - Jaipur
  - Kochi
  - Kolkata
  - Ludhiana
  - Mumbai
  - New Delhi
  - Pune
  - Vellore
- Italy (2):
  - Bologna, Emilia-Romagna
  - Udine, Friuli Venezia Giulia
- Riga, Latvia
- Lithuania (2):
  - Kaunas
  - Vilnius
- Malaysia (2):
  - George Town
  - Kuala Lumpur
- Monterrey, Mexico
- Peru (3):
  - Arequipa
  - Chiclayo
  - San Isidro
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Craiova (Dolj County)
- Russia (5):
  - Irkutsk
  - Kazan'
  - Krasnodar
  - Moscow
  - Saint Petersburg
- Singapore, Singapore
- Ljubljana, Slovenia
- Kiev, Ukraine
- United Kingdom (2):
  - London
  - Sutton

REFERENCES:
- [Derived] Propper D, Davidenko I, Bridgewater J, Kupcinskas L, Fittipaldo A, Hillenbach C, Klughammer B, Ducreux M. Phase II, randomized, biomarker identification trial (MARK) for erlotinib in patients with advanced pancreatic carcinoma. Ann Oncol. 2014 Jul;25(7):1384-1390. doi: 10.1093/annonc/mdu176. Epub 2014 May 14. PMID 24827134

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants with advanced pancreatic carcinoma with Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 to 2, who had failed 1 prior regimen of chemotherapy or who were considered unsuitable for chemotherapy, received placebo matching to erlotinib 150 mg tablet orally once daily until disease progression (PD), unacceptable toxicity, withdrawal, or death.
- Erlotinib: Participants with advanced pancreatic carcinoma with ECOG PS score of 0 to 2, who had failed 1 prior regimen of chemotherapy or who were considered unsuitable for chemotherapy, received erlotinib 150 mg orally once daily until PD, unacceptable toxicity, withdrawal, or death.
Period: Overall Study
Arm/Group | Placebo | Erlotinib
Started | 103 | 104
Switch to Open-Label Erlotinib | 57 (Participants with PD were given opportunity to switch.) | 0
Completed | 3 (Completed double-blind treatment.) | 2 (Completed double-blind treatment.)
Not Completed | 100 | 102
Not completed — Insufficient Therapeutic Response | 77 | 72
Not completed — Refused Treatment | 1 | 5
Not completed — Failure to Return | 1 | 0
Not completed — Adverse Event | 2 | 9
Not completed — Death | 19 | 15
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Erlotinib | Total
Number analyzed (Participants) | 103 | 104 | 207
Age, Customized [Number; unit: participants]
  Less than (<) 65 years | 72 | 62 | 134
  Greater than (>) 65 years | 31 | 42 | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 45 | 89
  Male | 59 | 59 | 118

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) was defined as the time from the date of randomization to the date of the first occurrence of PD or death whichever occurred first. Participants without event were censored at the date of last tumor assessment where non-progression was documented. Analysis was performed using Kaplan-Meier method.
Time Frame: From the time of randomization until progression of disease or death (up to 30 months)
Population: The Full-Analysis Set (FAS) was defined as all randomized patients. Participants were presented according to the therapy that they were randomized to receive.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 103 | 104
weeks | 5.9 [5.4 to 6.1] | 6.1 [5.9 to 6.4]
Statistical Analysis 1: Comparison: Placebo vs Erlotinib; Cox proportional hazards model was used to estimate the Hazard Ratio (erlotinib compared with placebo), including 95 percent (%) confidence intervals (CIs); Test type: Superiority or Other; p = 0.1909, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.63 to 1.10]

2. Secondary Outcome: Percentage of Participants With Best Overall Response Rate
Description: Response rate was defined as Complete Response (CR) or Partial Response (PR), according to response evaluation criteria in solid tumors (RECIST) Version 1.0 criteria, for at least 4 weeks at any time during randomized treatment (confirmed response). CR was defined as the disappearance of all target lesions. PR was defined as at least a 30% decrease in the sum of the longest diameters of target lesions.
Time Frame: From the time of randomization until progression of disease or death (up to 30 months)
Population: The FAS was defined as all randomized patients. Participants were presented according to the therapy that they were randomized to receive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 103 | 104
percentage of participants
  CR | 0 [0.0 to 3.5] | 0 [0.0 to 3.5]
  PR | 4 [1.1 to 9.6] | 1 [0.0 to 5.2]

3. Secondary Outcome: Percentage of Participants With Disease Control Rate (DCR)
Description: Disease control rates (DCR) were measured according to RECIST Version 1.0 criteria. Disease control was defined as being a responder or as having stable disease for at least 6 weeks post-randomization. Stable disease was defined as having neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease.
Time Frame: Randomization to Clinical Cutoff: 20 December 2010 (up to 30 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 103 | 104
percentage of participants | 19 [11.5 to 27.3] | 29 [19.5 to 37.5]

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of randomization to the date of death, regardless of the cause of death.
Time Frame: From the time of randomization until or death (up to 30 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 103 | 104
months | 3.1 [2.1 to 4.3] | 4.0 [2.8 to 4.8]

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who was administered a study treatment, regardless of whether or not the event had a causal relationship with the treatment. An AE, therefore, could be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the study treatment, whether or not related to the treatment.
Time Frame: Up to 28 days after discontinuation of study drug (up to 30 months)
Population: Safety population included all participants who received at least 1 dose of study medication and had a safety follow-up, whether withdrawn prematurely or not, were included in the safety population.
Measure: Number; unit: participants
Arm/Group | Placebo | Erlotinib
Number analyzed (Participants) | 103 | 104
participants | 71 | 90

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from baseline up to 28 days after discontinuation of study drug (up to 30 months)
Arm/Group | Placebo | Erlotinib
Serious Adverse Events (participants affected / at risk) | 11/103 | 21/104
Other Adverse Events (participants affected / at risk) | 70/103 | 81/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=103) | Erlotinib (N=104)
PYREXIA (General disorders) | 0 | 2
DEVICE OCCLUSION (General disorders) | 0 | 1
DRUG INTOLERANCE (General disorders) | 0 | 1
FATIGUE (General disorders) | 0 | 1
MUCOSAL INFLAMMATION (General disorders) | 1 | 0
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 | 1
BILIARY DILATATION (Hepatobiliary disorders) | 0 | 1
CHOLANGITIS (Hepatobiliary disorders) | 1 | 0
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 0 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 1
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYDROPNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
HAEMATEMESIS (Gastrointestinal disorders) | 1 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
BILIARY SEPSIS (Infections and infestations) | 0 | 2
MORGANELLA INFECTION (Infections and infestations) | 0 | 1
SEPSIS (Infections and infestations) | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 2
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
ANASTOMOTIC ULCER (Injury, poisoning and procedural complications) | 0 | 1
CONCUSSION (Injury, poisoning and procedural complications) | 1 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 0
VENOUS THROMBOSIS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=103) | Erlotinib (N=104)
DIARRHOEA (Gastrointestinal disorders) | 23 | 25
VOMITING (Gastrointestinal disorders) | 21 | 13
NAUSEA (Gastrointestinal disorders) | 10 | 22
ABDOMINAL PAIN (Gastrointestinal disorders) | 15 | 16
CONSTIPATION (Gastrointestinal disorders) | 17 | 8
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 12 | 10
ASCITES (Gastrointestinal disorders) | 9 | 1
RASH (Skin and subcutaneous tissue disorders) | 19 | 48
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 | 7
FATIGUE (General disorders) | 12 | 15
ASTHENIA (General disorders) | 7 | 12
PYREXIA (General disorders) | 7 | 12
MUCOSAL INFLAMMATION (General disorders) | 1 | 6
DECREASED APPETITE (Metabolism and nutrition disorders) | 13 | 18
ANAEMIA (Blood and lymphatic system disorders) | 8 | 11
WEIGHT DECREASED (Investigations) | 5 | 11
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 9 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 | 3
INSOMNIA (Psychiatric disorders) | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights